CLINICAL TRIAL: NCT00386516
Title: Phase 2, Multi-center, Open-label Trial to Evaluate Efficacy and Safety of GM-CT-01 in Combination With 5-FU as First Line Chemotherapy in Patients With Advanced Biliary Cancer
Brief Title: Study to Test the Benefit and Safety of GM-CT-01 in Combination With 5-FU to Treat Bile Duct and Gall Bladder Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Financing and re-organization
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAVFU-007
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2014-08

CONDITIONS: Cancer of the Bile Duct; Gallbladder Cancer
Keywords: cholangiocarcinoma; bile duct; biliary; intra-hepatic; extra-hepatic; gall bladder; cancer; carcinoma; metastatic; metastasis; advanced; recurrent
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Cholangiocarcinoma; Neoplasms; Carcinoma; Neoplasm Metastasis; Recurrence | interventions — galactomannan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GM-CT-01, 5-FU (Experimental): GM-CT-01 (280 mg/m2) combined with 5-FU (600 mg/m2) given 4 consecutive days in a 28 days cycle until disease progression.
  Interventions: Drug: GM-CT-01; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: GM-CT-01 — GM-CT-01 at 280 mg/m2 given IV for 4 consecutive days in 28 days cycle until disease progression
  Other Names: DAVANAT
Drug: 5-Fluorouracil — 5-FU given IV by infusion for 30, at 600 mg/m2 in combination with GM-CT-01 for 4 consecutive days in 28 days cycle until disease progression
  Other Names: 5-FU

SUMMARY:
The purpose of this clinical trial is to determine whether the combination of the established chemotherapeutic agent 5-fluorouracil(5-FU) and the large carbohydrate molecule GM-CT-01 is beneficial in treating advanced gall bladder and bile duct cancer.

DETAILED DESCRIPTION:
Determine the overall response rate (ORR) defined as complete response (CR)rate plus partial response (PR) rate using Response Evaluation Criteria in Solid Tumors (RECIST), as well as the stable disease (SD) rate in subjects with unresectable, locally advanced or metastatic cholangiocarcinoma or other biliary tract tumors treated with GM-CT-01 plus 5-Fluorouracil (DAVFU) at doses of 280 mg/m2 and 600 mg/m2, respectively, during cycles of 4 consecutive days of treatment followed by a 24-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Histologically or cytologically documented carcinoma primary to the intra- or extra-hepatic biliary system or gall bladder with clinical and/or radiologic evidence of unresectable, locally advanced or metastatic disease.
3. Prior neo-adjuvant or adjuvant therapy (including radiation therapy) is allowed provided it was completed at least 4 weeks before documented disease recurrence or metastasis.
4. Discontinuation of radiation therapy at least 3 weeks prior to Day 1 of Cycle 1. Radiation therapy will not be allowed while a subject is on study except for palliative radiation therapy to non-target lesions administered following consultation with the Medical Monitor.
5. Prior surgery must have been completed at least 14 days prior to Day 1 of Cycle 1.
6. Nne or more measurable target lesion(s) according to RECIST. Measurable lesion(s) must be outside of previous radiation field or demonstrate clear radiographic progression on serial imaging if within previous treatment field.
7. ECOG performance status less than or equal to 2.
8. Life expectancy greater or equal to 3 months.

Exclusion Criteria:

1. Central nervous system metastasis.
2. Bony metastasis as the sole metastasis.
3. Received prior chemotherapy or anti-angiogenesis agents including bevacizumab or erbitux or radiation therapy other than in a neo-adjuvant or adjuvant setting. No concomitant chemotherapy, anti-tumor biologic therapy, or radiation therapy is allowed.
4. If nitrosoureas or mitomycin C were used as neo-adjuvant or adjuvant therapy, then at least 6 weeks should have elapsed prior to treatment with DAVFU.
5. Active infection that requires treatment with systemic antibiotic, anti- fungal. or anti-viral therapy.
6. Congestive heart failure (Class III or IV in the NYHA functional classification system) or any other medical condition that would preclude the IV administration of up to approximately 200 mL of fluid over 30-60 minutes.
7. Unresolved biliary tract obstruction.
8. Known or clinically suspected infection with HIV.
9. Subject has a known intolerance to 5- FU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) defined as complete response (CR) rate plus partial response (PR) rate using Response Evaluation Criteria in Solid Tumors (RECIST) | When 18 valuable patients have completed 2nd CT
  A minimum of 18 subjects who meet the response evaluation criteria (per protocol population) will be enrolled in Stage 1. This require 2nd CT evaluation of tumor after minimum 2 cycles of treatments. CR, PR, SD and progressive disease (PD) as defined by RECIST criteria.
Stable disease (SD) rate and progression-free survival (PFS) times | When 18 valuable patients have completed 2nd CT
  A minimum of 18 subjects who meet the response evaluation criteria (per protocol population) will be enrolled in Stage 1. This require 2nd CT evaluation of tumor after minimum 2 cycles of treatments. SD and progressive disease (PD) as defined by RECIST criteria.

SECONDARY OUTCOMES:
Safety, tolerability and Quality of Life (QoL) | Any patient completed a drug treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Boston Medical Center, Boston, Massachusetts
  - University of Michigan, Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barrett Cancer Center, Cincinnati, Ohio